CLINICAL TRIAL: NCT03411005
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Lysine From Sorghum Protein, in Young Adult Men
Brief Title: Metabolic Availability of Lysine From Sorghum in Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Principal Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000058988
Record Dates: First submitted 2018-01-13; First posted 2018-01-25 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Healthy Men
Keywords: Lysine, Adult, Protein Quality

STUDY DESIGN:
Intervention Model Description: Each subject will randomly receive 3 levels of lysine provided as free amino acids, sorghum, or sorghum combined with lentils for a total of 8 studies x 3 days per study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic availability of lysine in Sorghum (Experimental): Participants will be seen initially for pre-study assessment (2 hour). They will then be studied at 8 levels of lysine intake.
  Subjects will visit SickKid's Clinical Research Center a total of 9 times, with each visit being at least one week before the next. All 9 visits must be made within 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein free-cookies and/or cooked sorghum with or without lentils, which will all be provided by the investigators.
  Interventions: Dietary Supplement: Metabolic availability of lysine in sorghum

INTERVENTIONS:
Dietary Supplement: Metabolic availability of lysine in sorghum — Four levels of lysine intakes will be provided by the reference protein drinks, 3 levels of lysine from sorghum and 1 level from sorghum with lentils.

SUMMARY:
Protein is the key determinant of growth and bodily functions. The quality of food proteins depend on their amino acid content and the amount of amino acids used by the body to make proteins. Globally Cereal Grains (CG) provide 50% of the calories and protein in the diet and exceed 80% in poorer developing countries. In many of those countries, sorghum is the major cereal grain in the diet. The protein in sorghum is low in the essential amino acid lysine. Hence sorghum protein is of low quality. Low lysine affects protein synthesis in the body. Cooking methods also affect the lysine available from foods to the body.The protein can be complemented by the addition of lentils to augment the low lysine content. However, lentils are prohibitively expensive in some developing countries.

As the human population increases, the world faces the continuous challenge of maximizing a limited food supply. Protein quality (PQ) evaluation of sorghum directly in humans would allow us to bridge the gap in knowledge between what is required and how best to provide.The information gathered from this project will provide the first direct experimental data on PQ of sorghum protein in humans on which nutrition recommendations can be built.

DETAILED DESCRIPTION:
Each subject will be part of 8 different experimental diets, and randomly assigned to one of the diets every time.

4 reference diet would be based on egg protein composition, 3 sorghum diets would have protein from cooked sorghum and 1 mixed meal would comprise of cooked sorghum and lentils.

Each experimental diet will be studied over 3 days: 2 adaptation and 1 study day. The 2 adaptation meals would be consumed at home. On the study day 3, following a 12-h overnight fast, subjects will come to the research unit at The Hospital for Sick Children, Toronto, ON for a period of 7.5 h and consume the diet as 9 hourly meals. The first 3 meals would be consumed at home.

For the duration of all experiments, subjects will consume a daily multivitamin supplement to ensure adequate vitamin intake.

Measurements:

Resting energy expenditure (REE) will be measured by open-circuit indirect calorimetry Body composition (fat and fat free mass) will be measured by BIA and Skin Fold. Breath samples will be collected after the 4th and 7th meals.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 - 49 yrs Healthy, with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes Stable Body Weight Not on any medications that could affect protein or amino acid metabolism e.g. steroids

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients)

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Assessment of the protein quality of Sorghum by determining the Metabolic availability of Lysine. | 2 years
  The MA of lysine in sorghum will be studied using the IAAO technique with L-(1-13C) phenylalanine as the indicator. In order to determine the MA of lysine, four levels of lysine will be tested; (5, 8, 12, 15 mg/kg/d which represent 13, 21, 32 and 40% of the lysine requirement for adults (37 mg/kg/d)) in five healthy adult men in a repeated measures design. Each subject will participate in 8 experiments: 4 lysine intakes as L-lysine from crystalline amino acid, 3 intakes of lysine from sorghum prepared by moist cooking and 1 experiment for dietary complementation with lentils. The MA of lysine will be estimated by comparing the IAAO response to varying intakes of Lysine in cooked sorghum compared with the IAAO response to lysine intakes in the reference protein (crystalline amino acid mixture patterned after egg protein) using the slope ratio method.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paoletti A, Fakiha A, Tul-Noor Z, Pencharz PB, Levesque CL, Ball RO, Kong D, Elango R, Courtney-Martin G. Bioavailable Lysine Assessed Using the Indicator Amino Acid Oxidation Method in Healthy Young Males is High when Sorghum is Cooked by a Moist Cooking Method. J Nutr. 2022 Mar 3;152(3):770-778. doi: 10.1093/jn/nxab410. PMID 34871427